CLINICAL TRIAL: NCT03262818
Title: Transvaginal Ultrasound and Photoacoustic Imaging of the Ovary
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201608016; 5R01CA151570-02 (NIH)
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Oophorectomy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transvaginal Ultrasound + Ultrasound/Photoacoustic imaging (Experimental): * Transvaginal ultrasound (US) prior to surgery
  * Immediately after the transvaginal US, US/PAI imaging will be performed
  * Once the surgeon has removed the ovary(ies) they will be imaged ex vivo. The in vivo and ex vivo US/PAI images will be compared with the final pathologic diagnosis
  Interventions: Device: Transvaginal ultrasound; Device: Ultrasound/Photoacoustic imaging

INTERVENTIONS:
Device: Transvaginal ultrasound — -Will be performed by US technologists at Washington University School of Medicine and read by Dr. Cary Siegel or Dr. Kathryn Robinson
  Other Names: Transvaginal US
Device: Ultrasound/Photoacoustic imaging — -The light illumination for the photoacoustic imaging system is provided by a wavelength-tunable Ti:Sapphire laser (LOTIS TII), optically pumped by an Nd:YAG laser (LOTIS TII) at 532 nm wavelength.
  Other Names: US/PAI

SUMMARY:
The investigators have developed co-registered photoacoustic and ultrasound (US) imaging technique that allows the investigators to visualize tumor structure and functional changes simultaneously, which may potentially reveal early tumor angiogenesis development that is not available by US alone. The ability to detect early angiogenesis changes, as well as tumor morphology changes in the ovary, using a non-invasive imaging modality will greatly enhance the care for women.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Referred to Washington University School of Medicine for conditions necessitating surgery to include at least a unilateral oophorectomy
* Willingness to participate in the study
* Able to provide informed consent

Exclusion Criteria

* Younger than 18 years of age
* Not able to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Measure PAI/ultrasound signatures from ovaries prior to surgery | Prior to surgery (no more than 30 days prior to surgery)
  -The transvaginal US will be performed by US technologists or radiologists at the Radiology Department and images will be read by one of the study radiologists either Dr. Cary Siegel or Dr. Kathryn Robinson of the Radiology Department. The reading will be categorized as normal, suspicious or highly suspicious. The scores will serve as a baseline comparison of US/PAI technique with the current clinical practice using US. Immediately after the transvaginal US, US/PAI imaging will be performed with the assistance of the US technologist or radiologist.

SECONDARY OUTCOMES:
Characterize the tissue images with pathologic diagnosis | At the time of surgery (no more than 30 days after PAI/US)
  -The in vivo and ex vivo PAI/US images with be compared with final pathologic diagnosis.
Refine the system and imaging algorithms based on the characteristic features of in vivo imaging | At the time of surgery (no more than 30 days after PAI/US)
  -Will be used to distinguish between benign and malignant ovarian tissues. Student t-test will be used for statistical significant test of each feature obtained from malignant and benign ovaries. Those features with p value less than 0.05 will be used as a predictor.

CONTACTS AND LOCATIONS:
Overall Officials: Cary L Siegel, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu